CLINICAL TRIAL: NCT05110157
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Valbenazine as Adjunctive Treatment in Subjects With Schizophrenia
Brief Title: Journey Study: Evaluate the Efficacy, Safety, and Tolerability of Valbenazine as Adjunctive Treatment for Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-ATS3019
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Valbenazine; Antipsychotic; VMAT2; NBI-98854; Dopamine; Journey; Neurocrine; PANSS; Adjunctive
MeSH Terms: conditions — Schizophrenia | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo once daily.
  Interventions: Drug: Placebo
- Vesicular monoamine transporter 2 (VMAT2) inhibitor (Experimental): Valbenazine once daily
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Placebo — Oral capsules
  Arms: Placebo
Drug: Valbenazine — Oral capsules
  Other Names: NBI-98854
  Arms: Vesicular monoamine transporter 2 (VMAT2) inhibitor

SUMMARY:
The primary objective for this study is to evaluate the effect of adjunctive valbenazine versus placebo on symptoms of schizophrenia in participants who have inadequate response to antipsychotic treatment.

DETAILED DESCRIPTION:
Phase 3, randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of valbenazine when administered orally once daily as adjunctive treatment in participants with schizophrenia who have had an inadequate response to antipsychotics. The study will enroll approximately 400 participants with a diagnosis of schizophrenia. The expected duration of study participation for each participant is approximately 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

• Participants must meet all of the following inclusion criteria:

1. Completed written informed consent.
2. At the time of signing the informed consent, participant must be ≥18 years of age
3. Medically confirmed diagnosis of schizophrenia as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
4. The initial diagnosis of schizophrenia must be ≥1 year before the screening visit.
5. Plasma levels for at least 1 of the participant's antipsychotic medications must be detectable by an available assay.
6. The participant is treated with a stable regimen antipsychotic medication.
7. Must meet all of the following criteria at the screening visit and Day 1:

   * PANSS total score ≥70
   * PANSS score of ≥4 on at least 1 of the following:

     * P1 (delusions)
     * P3 (hallucinations)
     * P6 (suspiciousness)
     * G9 (unusual thought content)
   * CGI-S score ≥4
   * Stable background antipsychotic medication dose between the screening visit and Day 1
   * Stable PANSS total score between the screening visit and Day 1
8. The participant is outpatient with stable symptomatology
9. The participant must have an adult informant (for example, a family member, relative, partner, social worker, caseworker, residential facility staff, or nurse).
10. Female participants of childbearing potential must agree to use contraception consistently from the screening visit until 30 days after the last dose of study drug or final study visit, whichever is longer.
11. Male participants must agree to use contraception consistently from screening until 30 days after last dose of study treatment.

Exclusion Criteria:

* Participants will be excluded from the study if they meet any of the following criteria:

  1. Pregnant or breastfeeding or plans to become pregnant during the study. This criterion must be reconfirmed prior to the first dose of study treatment on Day 1.
  2. Known hypersensitivity to any component of the formulation of valbenazine.
  3. Has history of treatment resistant schizophrenia.
  4. Evidence of depression as measured by a Calgary Depression Scale for Schizophrenia (CDSS) score ≥11 at the screening visit or Day 1.
  5. Participants with any suicidal behavior or suicidal ideation within 6 months before the screening visit or Day 1.
  6. Diagnosis of moderate or severe substance use disorder within the 6 months before the screening visit.
  7. Have a clinically significant unstable medical condition within 60 days before the screening visit in the judgement of the investigator or any laboratory value outside the normal range that is considered by the investigator to be clinically significant at the screening visit.
  8. Prior (within 6 months of the screening visit) or concomitant use of any VMAT2 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) total score from baseline to Week 10 | Baseline to week 10

SECONDARY OUTCOMES:
Change in Clinical Global Impression of Severity (CGI-S) score from baseline to Week 10 | Baseline to week 10
Change in Personal and Social Performance Scale (PSP) score from baseline to Week 10 | Baseline to week 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (74):
- United States (42):
  - Neurocrine Clinical Site, Phoenix, Arizona
  - Neurocrine Clinical Site, Rogers, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Bellflower, California
  - Neurocrine Clinical Site, Culver City, California
  - Neurocrine Clinical Site, Garden Grove, California
  - Neurocrine Clinical Site, Lemon Grove, California
  - Neurocrine Clinical Site, Long Beach, California
  - Neurocrine Clinical Site, Oceanside, California
  - Neurocrine Clinical Site, Pico Rivera, California
  - Neurocrine Clinical Site, Riverside, California
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, San Jose, California
  - Neurocrine Clinical Site, Santa Ana, California
  - Neurocrine Clinical Site, Stanford, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Aventura, Florida
  - Neurocrine Clinical Site, Coral Gables, Florida
  - Neurocrine Clinical Site, Daytona Beach, Florida
  - Neurocrine Clinical Site, Hialeah, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Miami Lakes, Florida
  - Neurocrine Clinical Site, Okeechobee, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, West Palm Beach, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Evanston, Illinois
  - Neurocrine Clinical Site, Springfield, Illinois
  - Neurocrine Clinical Site, Grand Rapids, Michigan
  - Neurocrine Clinical Site, St Louis, Missouri
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Las Vegas, Nevada
  - Neurocrine Clinical Site, Cedarhurst, New York
  - Neurocrine Clinical Sites, Glen Oaks, New York
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, Charlotte, North Carolina
  - Neurocrine Clinical Site, Dayton, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Austin, Texas
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, Houston, Texas
- Argentina (2):
  - Neurocrine Clinical Site, Buenos Aires
  - Neurocrine Clinical Site, Córdoba
- Bulgaria (13):
  - Neurocrine Clinical Site, Kardzhali
  - Neurocrine Clinical Site, Lovech
  - Neurocrine Clinical Site 1, Pleven
  - Neurocrine Clinical Site 2, Pleven
  - Neurocrine Clinical Site 1, Plovdiv
  - Neurocrine Clinical Site 2, Plovdiv
  - Neurocrine Clinical Site, Plovdiv
  - Neurocrine Clinical Site, Rousse
  - Neurocrine Clinical Site 1, Sofia
  - Neurocrine Clinical Site 2, Sofia
  - Neurocrine Clinical Site, Sofia
  - Neurocrine Clinical Site, Veliko Tarnovo
  - Neurocrine Clinical Site, Vratsa
- Serbia (17):
  - Neurocrine Clinical Site 1, Belgrade
  - Neurocrine Clinical Site 2, Belgrade
  - Neurocrine Clinical Site 3, Belgrade
  - Neurocrine Clinical Site 4, Belgrade
  - Neurocrine Clinical Site 5, Belgrade
  - Neurocrine Clinical Site 6, Belgrade
  - Neurocrine Clinical Site, Belgrade
  - Neurocrine Clinical Site, Gornja Toponica
  - Neurocrine Clinical Site 1, Kovin
  - Neurocrine Clinical Site 2, Kovin
  - Neurocrine Clinical Site 1, Kragujevac
  - Neurocrine Clinical Site 2, Kragujevac
  - Neurocrine Clinical Site 3, Kragujevac
  - Neurocrine Clinical Site, Niš
  - Neurocrine Clinical Site, Novi Kneževac
  - Neurocrine Clinical Site, Vojvodina
  - Neurocrine Clinical Site, Vršac

IPD SHARING:
Plan to Share IPD: No